CLINICAL TRIAL: NCT04893486
Title: A Multicenter, Phase 2B, Randomized, Double-Blind, Stratified, Vehicle-Controlled Study Evaluating The Safety And Efficacy Of QTORIN 3.9% Sirolimus Topical Gel In Prevention Of BCCs In Patients With Gorlin Syndrome
Brief Title: CODY: A Study Evaluating The Safety And Efficacy Of QTORIN 3.9% Sirolimus Topical Gel For The Prevention Of Basal Cell Carcinomas (BCCs) In Patients With Gorlin Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palvella Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PALV-04
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: BCCs in Gorlin Syndrome Patients
Keywords: Gorlin Syndrome; Basal Cell Carcinoma; Nevoid basal cell carcinoma syndrome; Basal cell nevus syndrome BCNS; Gorlin Syndrome Alliance; Prevention; Topical; Sirolimus
MeSH Terms: conditions — Basal Cell Nevus Syndrome; Carcinoma, Basal Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: PTX-022
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle comparator

INTERVENTIONS:
Drug: PTX-022 — QTORIN 3.9 % Sirolimus Topical Gel
  Arms: Active
Drug: Vehicle comparator — Vehicle comparator topical gel
  Arms: Vehicle

SUMMARY:
A Phase 2b study looks at the safety and efficacy of a treatment that is being investigated for people with certain diseases. This study will be conducted at multiple centers in the United States where participants with Gorlin Syndrome, also known as basal cell nevus syndrome, will be randomly placed into two groups; one group will receive the active topical gel, the other a topical vehicle gel, also know as placebo. Participants will apply this topical product to their face once a day for 6 months. The study will be looking at the number of new BCCs that develop on the faces of all the participants during this time.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults, 18 years or older
* Meet diagnostic criteria for Gorlin Syndrome
* Willing to avoid application of a non-study topical medication to the face (prescription or over the counter) during the study.
* Willing to forego treatment of BCCs with anything other than the study medication except when the Investigator believes that delay of treatment of a BCC potentially might compromise the health of the subject. During the trial, the only allowed form of BCC treatment is surgical.
* Participant will be encouraged to use their preferred sunscreen with a sun protector factor (SPF) of at least 30 daily

Key Exclusion Criteria:

* Recently participated in a clinical trial evaluating an investigational product for the treatment of BCCs or Gorlin Syndrome within 3 months prior to to starting study medication. Participant can start the study screening period prior to completing the 3 month washout.
* Recently used topical or systemic (oral) treatment that might interfere with the evaluation of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Number of new biopsy confirmed BCCs that develop on the face compared between the active and vehicle treatment arms | Month 6
Incidence of dermatological, treatment emergent adverse events after treatment with active | Month 6

SECONDARY OUTCOMES:
Percentage of participants developing 2 or more new biopsy confirmed BCCs on the face. | Month 6
Percentage of participants developing 1 or more new biopsy confirmed BCCs on the face. | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: David Bickers, MD, Study Chair — Columbia University; Joyce Teng, MD, Principal Investigator — Stanford University
Locations (16):
- United States (14):
  - Mayo Clinic, Scottsdale, Arizona
  - Burke Pharmaceuticals Research, Hot Springs, Arkansas
  - Stanford Univeristy, Palo Alto, California
  - Park Avenue Dermatology, Orange Park, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Gwinett Clinical Research Center, Snellville, Georgia
  - Clinical Coordinating Center (Minnesota), New Brighton, Minnesota
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - DermResearch Inc, Austin, Texas
  - University of Utah, Murray, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- United Kingdom (2):
  - St. Pancras Clinical Research, London
  - Salford Foundation Trust, Salford

REFERENCES:
- See also: Sign-up to be contacted about participation in the clinical trial — http://weblink.donorperfect.com/clinicaltrialinterest
- See also: Gorlin Syndrome Alliance — http://gorlinsyndrome.org/